CLINICAL TRIAL: NCT00397657
Title: ARBITER 6: ARterial Biology for the Investigation of the Treatment Effects of Reducing Cholesterol 6 - HDL and LDL Treatment Strategies in Atherosclerosis (HALTS)
Brief Title: Comparative Study of the Effect of Ezetimibe Versus Extended-Release Niacin on Atherosclerosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Independent steering committee has stopped the trial based on results of a prespecified, blinded interim analysis. It was not stopped due to safety concerns.
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Abbott (Industry)
Responsible Party: Allen J Taylor, MD, Medstar Research Institute and Washington Hospital Center, Washington DC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-12027
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Atherosclerosis
Keywords: carotid intima media thickness; atherosclerosis; niacin; coronary heart disease; HDL-C; LDL-C
MeSH Terms: conditions — Atherosclerosis; Coronary Disease | interventions — Ezetimibe

ARMS (2):
- Extended release niacin (Active Comparator)
  Interventions: Drug: extended release niacin; Drug: ezetimibe
- Ezetimibe (Active Comparator)
  Interventions: Drug: ezetimibe

INTERVENTIONS:
Drug: extended release niacin — Extended release niacin will be started at 1000mg and titrated to 2000mg once a day
  Arms: Extended release niacin
Drug: ezetimibe — Ezetimibe 10mg once daily

SUMMARY:
Recent evidence on the use of statin therapy indicates the potential for ultra-low levels of low-density lipoprotein (LDL-C) to provide greater protection from recurrent coronary heart disease (CHD) events. Thus, in August 2005, the guidelines for the treatment of lipid disorders (NCEP ATPIII) were revised to indicate that an LDL-C treatment goal of 70 mg/dL (revised from 100 mg/dL) was optional for patients with known CHD. In these same guidelines, low levels of high-density lipoprotein (HDL-C) are also suggested but not specifically proscribed as a target of therapy. Recently the ARBITER 2 trial has provided the first evidence of the potential of raising HDL-C with extended release niacin when added to statin monotherapy. However, whether this approach would be superior to a strategy in which lower concentrations of LDL-C are targeted is unknown.

The purpose of ARBITER 6 - HALTS is to compare HDL and LDL-focused strategies of lipid treatments for their effects of atherosclerosis. This study is a prospective, randomized, open-label, blinded endpoint trial comparing treatment strategies of either HDL-raising therapies or LDL reduction for dyslipidemia on carotid atherosclerosis. Subjects with known atherosclerotic coronary or vascular disease or otherwise at high cardiovascular risk through the presence of a coronary risk equivalent who are currently being treated with a statin will be eligible. Subjects will be randomly assigned in an allocation-concealed fashion to open label treatment with either Ezetimibe 10 mg/d for additional LDL-lowering OR Extended-release niacin (1 gm/d, titrated to max tolerable dose up to 2 gm/d) for HDL improvement.

The effects of these 2 different strategies of intensified lipid management on atherosclerosis will be assessed by the change in the carotid intima-media thickness, a validated surrogate endpoint. The data will help guide clinicians on the potential benefits of these lipid treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ≥ 30 years old with either known atherosclerotic coronary or vascular disease OR coronary risk equivalents defined as either:

  * diabetes mellitus,
  * multiple coronary risk factors with a Framingham Risk Score > 2% per year, or
  * an elevated coronary calcium score (> 400 for men, > 200 for women)
* Currently being treated with a statin (Simvastatin 20 mg/d or its equivalent) as monotherapy for treatment of hyperlipidemia
* Recent lipids (within the past 3 months without interval change in the statin regimen) showing both: LDL-C < 100 mg/dL and HDL-C < 50 mg/dL (men) or < 55 mg/dL (women)

Exclusion Criteria:

* Current use of or known intolerance to niacin or ezetimibe
* Known history of liver disease (cirrhosis, chronic hepatitis) or abnormal liver associated enzymes, > 3x the upper laboratory reference value
* Enrollment in another drug or device research protocol
* Females who are pregnant, expect to get pregnant during the course of the study, or are breastfeeding

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-08 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the change in carotid intima-media thickness between groups after 14 months | 14 months

SECONDARY OUTCOMES:
The change in lipid values and lipid subfractions | 14 months
A composite endpoint consisting of all major adverse cardiovascular events (coronary heart disease death, myocardial infarction, myocardial revascularization, admission to the hospital for an acute coronary syndrome) | 14 months
Drug discontinuation due to adverse effects | 14 months
Quality of life measured with the EQ-5D questionnaire- a generic questionnaire for describing and valuing subjects' health-related quality of life that has been studied in cardiovascular subjects | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Allen J Taylor, MD, Principal Investigator — Medstar Research Institute and Washington Hospital Center, Washington DC.
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Washington Adventist Hospital, Takoma Park, Maryland

REFERENCES:
- [Background] Cashin-Hemphill L, Mack WJ, Pogoda JM, Sanmarco ME, Azen SP, Blankenhorn DH. Beneficial effects of colestipol-niacin on coronary atherosclerosis. A 4-year follow-up. JAMA. 1990 Dec 19;264(23):3013-7. PMID 2243429
- [Background] Mack WJ, Selzer RH, Hodis HN, Erickson JK, Liu CR, Liu CH, Crawford DW, Blankenhorn DH. One-year reduction and longitudinal analysis of carotid intima-media thickness associated with colestipol/niacin therapy. Stroke. 1993 Dec;24(12):1779-83. doi: 10.1161/01.str.24.12.1779. PMID 8248954
- [Background] Brown G, Albers JJ, Fisher LD, Schaefer SM, Lin JT, Kaplan C, Zhao XQ, Bisson BD, Fitzpatrick VF, Dodge HT. Regression of coronary artery disease as a result of intensive lipid-lowering therapy in men with high levels of apolipoprotein B. N Engl J Med. 1990 Nov 8;323(19):1289-98. doi: 10.1056/NEJM199011083231901. PMID 2215615
- [Background] Azen SP, Mack WJ, Cashin-Hemphill L, LaBree L, Shircore AM, Selzer RH, Blankenhorn DH, Hodis HN. Progression of coronary artery disease predicts clinical coronary events. Long-term follow-up from the Cholesterol Lowering Atherosclerosis Study. Circulation. 1996 Jan 1;93(1):34-41. doi: 10.1161/01.cir.93.1.34. PMID 8616937
- [Background] Brown BG, Zhao XQ, Chait A, Fisher LD, Cheung MC, Morse JS, Dowdy AA, Marino EK, Bolson EL, Alaupovic P, Frohlich J, Albers JJ. Simvastatin and niacin, antioxidant vitamins, or the combination for the prevention of coronary disease. N Engl J Med. 2001 Nov 29;345(22):1583-92. doi: 10.1056/NEJMoa011090. PMID 11757504
- [Background] Taylor AJ, Sullenberger LE, Lee HJ, Lee JK, Grace KA. Arterial Biology for the Investigation of the Treatment Effects of Reducing Cholesterol (ARBITER) 2: a double-blind, placebo-controlled study of extended-release niacin on atherosclerosis progression in secondary prevention patients treated with statins. Circulation. 2004 Dec 7;110(23):3512-7. doi: 10.1161/01.CIR.0000148955.19792.8D. Epub 2004 Nov 10. PMID 15537681
- [Background] Nissen SE, Tuzcu EM, Schoenhagen P, Brown BG, Ganz P, Vogel RA, Crowe T, Howard G, Cooper CJ, Brodie B, Grines CL, DeMaria AN; REVERSAL Investigators. Effect of intensive compared with moderate lipid-lowering therapy on progression of coronary atherosclerosis: a randomized controlled trial. JAMA. 2004 Mar 3;291(9):1071-80. doi: 10.1001/jama.291.9.1071. PMID 14996776
- [Background] Taylor AJ, Kent SM, Flaherty PJ, Coyle LC, Markwood TT, Vernalis MN. ARBITER: Arterial Biology for the Investigation of the Treatment Effects of Reducing Cholesterol: a randomized trial comparing the effects of atorvastatin and pravastatin on carotid intima medial thickness. Circulation. 2002 Oct 15;106(16):2055-60. doi: 10.1161/01.cir.0000034508.55617.65. PMID 12379573
- [Background] Davidson MH, McGarry T, Bettis R, Melani L, Lipka LJ, LeBeaut AP, Suresh R, Sun S, Veltri EP. Ezetimibe coadministered with simvastatin in patients with primary hypercholesterolemia. J Am Coll Cardiol. 2002 Dec 18;40(12):2125-34. doi: 10.1016/s0735-1097(02)02610-4. PMID 12505224
- [Background] Burke GL, Evans GW, Riley WA, Sharrett AR, Howard G, Barnes RW, Rosamond W, Crow RS, Rautaharju PM, Heiss G. Arterial wall thickness is associated with prevalent cardiovascular disease in middle-aged adults. The Atherosclerosis Risk in Communities (ARIC) Study. Stroke. 1995 Mar;26(3):386-91. doi: 10.1161/01.str.26.3.386. PMID 7886711
- [Background] Jukema JW, Bruschke AV, van Boven AJ, Reiber JH, Bal ET, Zwinderman AH, Jansen H, Boerma GJ, van Rappard FM, Lie KI, et al. Effects of lipid lowering by pravastatin on progression and regression of coronary artery disease in symptomatic men with normal to moderately elevated serum cholesterol levels. The Regression Growth Evaluation Statin Study (REGRESS). Circulation. 1995 May 15;91(10):2528-40. doi: 10.1161/01.cir.91.10.2528. PMID 7743614
- [Background] Taylor AJ, Lee HJ, Sullenberger LE. The effect of 24 months of combination statin and extended-release niacin on carotid intima-media thickness: ARBITER 3. Curr Med Res Opin. 2006 Nov;22(11):2243-50. doi: 10.1185/030079906x148508. PMID 17076985
- [Derived] Taylor AJ, Villines TC, Stanek EJ. Paradoxical progression of atherosclerosis related to low-density lipoprotein reduction and exposure to ezetimibe. Eur Heart J. 2012 Dec;33(23):2939-45. doi: 10.1093/eurheartj/ehs105. Epub 2012 May 7. PMID 22564353
- [Derived] Villines TC, Stanek EJ, Devine PJ, Turco M, Miller M, Weissman NJ, Griffen L, Taylor AJ. The ARBITER 6-HALTS Trial (Arterial Biology for the Investigation of the Treatment Effects of Reducing Cholesterol 6-HDL and LDL Treatment Strategies in Atherosclerosis): final results and the impact of medication adherence, dose, and treatment duration. J Am Coll Cardiol. 2010 Jun 15;55(24):2721-6. doi: 10.1016/j.jacc.2010.03.017. PMID 20399059
- [Derived] Taylor AJ, Villines TC, Stanek EJ, Devine PJ, Griffen L, Miller M, Weissman NJ, Turco M. Extended-release niacin or ezetimibe and carotid intima-media thickness. N Engl J Med. 2009 Nov 26;361(22):2113-22. doi: 10.1056/NEJMoa0907569. Epub 2009 Nov 15. PMID 19915217